CLINICAL TRIAL: NCT05182606
Title: Consensus-based Algorithms to Address Opioid Misuse Behaviors Among Individuals Prescribed Long-term Opioid Therapy: Developing Implementation Strategies and Pilot Testing
Brief Title: Consensus-based Algorithms to Address Opioid Misuse Behaviors Among Individuals Prescribed Long-term Opioid Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jessica Merlin, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20030189; R34DA050004 (NIH)
Record Dates: First submitted 2021-11-28; First posted 2022-01-10 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Opioid Misuse; Chronic Pain
Keywords: Long-Term Opioid Therapy; Algorithms; Opioid Misuse; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Investigators will conduct a pilot trial to assess the feasibility, acceptability, and preliminary effectiveness of the Algorithm Implementation Package across three University of Pittsburgh Medical Center (UPMC) primary care practices. The intervention will be implemented using a staggered rollout across the three clinics - General Internal Medicine Oakland will receive the intervention first, followed by Northern Medical Associates Hampton and Wexford. All clinics will receive the same intervention. Feasibility and acceptability will be assessed once only after the 6- or 9-month implementation period through clinician surveys and qualitative interviews. Preliminary effectiveness will be evaluated using electronic health record (EHR) data assessing reductions in concerning opioid-related behaviors and increases in the diagnosis and treatment of Opioid Use Disorder.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation Bundle (Experimental): The 'Implementation Bundle' was integrated into all three participating clinics over six to nine months.
  Interventions: Behavioral: Pilot study of algorithms implementation package

INTERVENTIONS:
Behavioral: Pilot study of algorithms implementation package — The algorithm implementation package includes a link to the algorithms in the Electronic Health Record, Smartphrases, audited feedback, and instructions.

SUMMARY:
The NIH Helping to End Addiction Long-term (HEAL) initiative has identified a critical next step to addressing the opioid crisis: improving treatments for opioid misuse behaviors (e.g., using more opioids than prescribed, illicit substance use) in patients prescribed long-term opioid therapy for chronic pain. In previous work, the investigators have developed innovative consensus-based algorithms to manage these behaviors. By developing implementation strategies for these algorithms, this project is directly responsive to the HEAL initiative and promises to reduce opioid misuse-related harms.

DETAILED DESCRIPTION:
Despite a growing understanding of the risks of long-term opioid therapy (LTOT), it continues to be frequently prescribed and remains a mainstay of treatment for chronic pain. The Centers for Disease and Control (CDC) Guideline for Prescribing Opioids for Chronic Pain is geared toward primary care providers and has been adopted as the standard of care by many healthcare organizations and insurers. Importantly, it encourages monitoring of patients on LTOT for opioid-related harms. By implementing monitoring, primary care providers may uncover various concerning behaviors, sometimes called aberrant drug-related behaviors or opioid misuse behaviors, that arise among individuals prescribed LTOT for chronic pain. These behaviors (e.g., missed appointments, using more opioid medication than prescribed, asking for an increase in opioid dose, aggressive behavior, and alcohol and other substance use) are common, concerning, and may represent unsafe use of LTOT or a developing opioid use disorder (OUD). However, the CDC Guideline and other existing evidence do not provide specific, detailed guidance about how to address concerning behaviors when they occur. Therefore, there is a critical need to understand how to best respond to these behaviors. The long-term goal of our program of research is to reduce LTOT-related harms, particularly from opioid misuse, and diminish their impact on the U.S. opioid epidemic. As a first step toward accomplishing this goal, the investigators conducted a Delphi study to rigorously establish consensus-based approaches to managing common and challenging concerning behaviors, from which algorithms were created. Identifying and operationalizing implementation strategies using an evidence-based framework are the critical next steps that must occur before any testing of the algorithms.

The investigators successfully uncovered optimal implementation strategies through primary care provider experiences with Standardized Patients (SPs) followed by Consolidated Framework for Implementation Research (CFIR)- and Expert Recommendations for Implementing Change (ERIC)-guided individual interviews. Using our prior expertise developing clinic-wide opioid risk reduction strategies and a Patient-Provider advisory board, the investigators developed a comprehensive "implementation package" that can be delivered to primary care practices.

The investigators now aim to conduct a pilot trial to test the algorithm implementation package. Guided by the CFIR-based implementation plan and using the implementation package that the investigators developed, pilot trial will be conducted to investigate feasibility, acceptability, and preliminary effectiveness of the algorithm implementation package.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians practicing at UPMC community primary care clinics.

Exclusion Criteria:

* Clinicians not practicing at UPMC community primary care clinics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Merlin, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three University of Pittsburgh Medical Center (UPMC) clinics were recruited for the study, with clinicians at these clinics participating in the implementation. The toolkit was sequentially integrated into the practices between September 2022 and September 2023.
Pre-assignment Details: We reduced our sample to 3 clinics: two community with the same director, and one larger academic practice. We started the intervention at the academic clinic 2 months before the two community clinics for logistical reasons. Because not all physicians reported information about clinic affiliation, data are presented into a single arm. The academic clinic implementation lasted 6 months and the two community clinics 9 months. All 3 clinics were assessed 12 months pre- and post-implementation.
Units Other Than Participants: clinics
Groups:
- Implementation Bundle: The 'Implementation Bundle' was integrated into participating clinics over six or nine months. This algorithm implementation package included a link to the algorithms in the Electronic Health Record, Smartphrases, audited feedback, and instructions.
Period: Pre-implementation (12 Months Before)
Arm/Group | Implementation Bundle
Started | 49; 3 clinics
Completed | 49; 3 clinics
Not Completed | 0; 0 clinics
Period: Implementation
Arm/Group | Implementation Bundle
Started | 49; 3 clinics
Completed | 49; 3 clinics
Not Completed | 0; 0 clinics
Period: Post-implementation (12 Months After)
Arm/Group | Implementation Bundle
Started | 49; 3 clinics
Completed | 20; 3 clinics
Not Completed | 29; 0 clinics
Not completed — Did not participate in the post-implementation survey | 29

BASELINE CHARACTERISTICS:
Groups:
- Implementation Bundle: The 'Implementation Bundle' was integrated into participating clinics over six to nine months. This algorithm implementation package included a link to the algorithms in the Electronic Health Record, Smartphrases, audited feedback, and instructions.
Arm/Group | Implementation Bundle
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 49
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49
Provider at UPMC [Count of Participants; unit: Participants] | 49

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Algorithms
Description: The number of algorithms used by physicians was assessed via a survey administered at the end of the 6- or 9-month implementation period, measuring self-reported toolkit utilization during the study. Our primary feasibility benchmark will be that 80% of physicians report using at least one algorithm during the study period.
Time Frame: At the end of the 6- or 9-month implementation period
Population: Physicians from the three participating clinics who agreed to participate in the post-implementation survey.
Measure: Count of Participants; unit: Participants
Groups:
- Implementation Bundle: The 'Implementation Bundle' was integrated into participating clinics over 6-9 months. This algorithm implementation package included a link to the algorithms in the Electronic Health Record, Smartphrases, audited feedback, and instructions.
Arm/Group | Implementation Bundle
Number analyzed (Participants) | 20
Participants
  Physicians who used at least one algorithm | 7
  Physicians who did not use any algorithm or did not respond to this question | 13

2. Primary Outcome: Acceptability of Algorithms
Description: Acceptability of the algorithms was assessed via a self-report survey administered at the end of the 6- or 9-month implementation period, measuring physicians' awareness of the algorithms and self-reported toolkit use within six months of implementation. Our primary acceptability benchmark is that at least 80% of physicians report awareness of the algorithm implementation and at least 50% report using the algorithms during the study period. Additionally, qualitative interviews with physicians and staff provided further insights, which were analyzed using thematic analysis.
Time Frame: At the end of the 6- or 9-month implementation period
Population: Physicians from the three participating clinics who agreed to participate in post-implementation surveys.
Measure: Count of Participants; unit: Participants
Groups:
- Implementation Bundle: The 'Implementation Bundle' was integrated into participating clinics over six months. This algorithm implementation package included a link to the algorithms in the Electronic Health Record, Smartphrases, audited feedback, and instructions.
Arm/Group | Implementation Bundle
Number analyzed (Participants) | 20
Participants
  Physicians aware of algorithm implementation | 19
  Physicians who used at least one algorithm | 7

3. Secondary Outcome: Preliminary Effectiveness of Algorithms - MME Reduction ≥10%
Description: Number of long-term opioid therapy (LTOT) patients whose 90-day average Morphine Milligram Equivalents (MME) decreased at or above a margin of 10% from the start of the reporting period to the end of the reporting period.
Time Frame: Pre-implementation (12 months), implementation (6 to 9 months), post-implementation (12 months)
Population: Outcome values are aggregated from electronic health records (EHR) for LTOT patients attributed to participating physicians (n=49). Patients EHRs contributed outcome data but were not enrolled study participants. Number of LTOT patients whose 90-day average MMEs decreased at or above a margin of 10% from the start of the reporting period to the end of the reporting period.
Measure: Number; unit: Clinic patients
Arm/Group | Implementation Bundle
Number analyzed (Participants) | 49
Clinic patients
  Pre-implementation Period | 297
  Implementation Period | 122
  Post-implementation Period | 270

4. Secondary Outcome: Preliminary Effectiveness - Average MME Within Last 90 Days
Description: Average morphine milligram equivalents (MME) among long-term opioid therapy (LTOT) patients during the last 90 days of each period.
Time Frame: Pre-implementation (12 months), implementation (6 or 9 months), post-implementation (12 months)
Population: Outcome values are aggregated from electronic health record (EHR) data for LTOT patients attributed to participating physicians (n=49). Patient EHR data contributed to the outcomes, but patients were not enrolled as study participants. Row values reflect patient-level means (SD) by period. Means aggregate monthly 90-day MME within each period.
Measure: Mean (Standard Deviation); unit: 90-day average MME (mg/day)
Arm/Group | Implementation Bundle
Number analyzed (Participants) | 49
90-day average MME (mg/day)
  Pre-implementation Period | 105.25 (16.27)
  Implementation Period | 96.76 (21.06)
  Post-implementation Period | 96.48 (16.34)

5. Secondary Outcome: Preliminary Effectiveness of Algorithms - Opioid Discontinuation
Description: Number of long-term opioid therapy (LTOT) patients whose 90-day average Morphine Milligram Equivalents (MME) at the start of this reporting period was 0.
Time Frame: Pre-implementation (12 months), implementation (6 to 9 months), post-implementation (12 months)
Population: Outcome values are aggregated from electronic health records (EHR) for LTOT patients attributed to participating physicians (n=49). Patients EHRs contributed outcome data but were not enrolled study participants. Row values reflect patient-level totals by period.
Measure: Number; unit: Clinic patients
Arm/Group | Implementation Bundle
Number analyzed (Participants) | 49
Clinic patients
  Pre-implementation Period | 95
  Implementation Period | 109
  Post-implementation Period | 166

6. Secondary Outcome: Preliminary Effectiveness of the Algorithms - New OUD Diagnoses
Description: New opioid use disorder (OUD) diagnoses documented in the electronic health record (EHR) among all patients seen by participating physicians, by period. No new OUD diagnoses were documented in any period.
Time Frame: Pre-implementation (12 months), implementation (6 to 9 months), post-implementation (12 months)
Population: as for outcome 5
Measure: Number; unit: Diagnoses
Arm/Group | Implementation Bundle
Number analyzed (Participants) | 49
Diagnoses
  Pre-implementation period | 0
  Implementation period | 0
  Post-implementation period | 0

ADVERSE EVENTS:
Time Frame: 18 months for the academic clinic, 21 months for the two community clinics
Description: Although we are using electronic health record (EHR) data from the pre-implementation period for comparison purposes, these data were extracted retrospectively after the implementation phase. Because no active intervention was in place during the pre-implementation phase, adverse events cannot be collected for that period.
Groups:
- Implementation: The 'Implementation Bundle' was integrated into participating clinics over a staggered 6-9 month period. The algorithm implementation package included a link to the algorithms in the Electronic Health Record, Smartphrases, audited feedback, and instructions. The academic clinic began implementation two months prior to the two community-based clinics.
- Post-implementation: This period reflects the 12 months following the active implementation phase. During this time, clinics retained access to the algorithm tools, but no additional implementation support was provided. This period was used to assess maintenance of algorithm use.
Arm/Group | Implementation | Post-implementation
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

LIMITATIONS AND CAVEATS:
The study's findings are limited by its pilot nature, focusing on a small number of clinics and clinicians. Results may not be generalizable to other settings or populations. Additionally, qualitative data were collected from a subset of participants, which may not fully represent all perspectives. The limited follow-up time may also restrict the interpretation of longer-term outcomes or broader feasibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT05182606/Prot_SAP_000.pdf